CLINICAL TRIAL: NCT02211703
Title: National Epidemiologic Survey on the Incidence of Perioperative Hypothermia in Patients With Elective Surgery Under General Anesthesia in China
Brief Title: National Epidemiologic Survey on the Incidence of Perioperative Hypothermia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Jie YI (Other)
Collaborators: Medical Consulting Center (Network)
Responsible Party: Sponsor-Investigator, Jie YI, Associate Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: MDI0091
Record Dates: First submitted 2014-08-06; First posted 2014-08-07 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-08

CONDITIONS: Hypothermia
Keywords: perioperative hypothermia; Epidemiology; Tympanic temperature
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation: This is an epidemiology study in which all the data from the subjects enrolled will be collected and analysis to investigate the current patient warming condition and actual perioperative hyperthermia rate in the elective operation with general anesthesia. During the whole procedure none intervention is administered.

SUMMARY:
Study Objective:

* to project the incidence of perioperative hypothermia in patients with elective surgery under general anesthesia in China
* to determine the risk factors associated with perioperative hypothermia.
* to explore the patient outcome of hypothermia such as cardiovascular events, wound infection,hospital stay and so on.

Study Design: The present study is a cross-sectional study with 30-day follow-up period.

DETAILED DESCRIPTION:
This survey was anticipated to enroll 2208 patients with elective surgery under general anesthesia from 28 hospitals or so in China. After obtaining approval from the Ethical Committee related to research involving human subjects,the investigators will enroll the patients according to the inclusion and exclusion criterion. The tympanic temperature will be monitored at the following time points respectively: Arriving at waiting area, entering the OR room, 5 min before and after anesthesia induction, every 15 min during the operation, after 2h the tympanic temperature will be monitored at every 30 min, Tympanic temperature will also be taken when the surgery complete and when patients arrived at PACU. Other information will also be collected including the type and dosage of anesthesia drug,duration of surgery and anesthesia, patient warming method，operation room temperature, the amount of the infusion of intravenous fluids and blood and their warming techniques during the whole operation procedure. The postoperative follow-up will be conducted and recorded within 30 days after operation(for implantation surgery, the follow-up will be conducted within 90 days postoperatively ) which includes ICU stays, hospital stays, wound infection, new cardiovascular events.etc.

The contract research organization will be delegated to do an on site monitor once a month (online monitor once a week) for each hospital participate the survey during the recruitment and perform the source data validation at the same time to review the related medical records,source data and the case report forms, etc.to ensure the data accuracy and completeness.

Data management will be conducted through the whole survey procedure. In order to guarantee the validation of the data, two data managing staffs will input and verify the data independently.

Statistical analysis software (SAS9.2) was used for the calculation of all the statistical analyses. The number of cases, mean, standard deviation, median value, maximal value and minimal value should be calculated for the descriptions of the qualitative parameters. Number of cases and percentages are used for the descriptions on the classification parameters.Two side test is used for all the statistical tests, P<0.05 indicates that the difference is statistically significant (unless indicated otherwise), and 95% confidence is used as the confidence interval.

ELIGIBILITY:
Inclusion Criteria:

* Male or female，age≥18 Subjects will undergo an elective surgeries with general anaesthesia The duration of operation is expected to be over 60 minutes The subjects agreed to participate in the study and signed the consent form.

Exclusion Criteria:

* Central high fever, including that induced by cerebrovascular, disease, cerebral trauma, cerebral, surgeries, epilepsy and acute hydrocephalus Thermoregulation abnormalities including malignant hyperthermia (MHS) and neuroleptic malignant syndrome Hypothyroidism or hyperthyroidism diagnosed by substantial evidence Infectious fever Temperature is higher than 37.8℃ within 3 days before surgery Diseases or surgery that may lead to inaccuracy in measurement of era thermometer , such as ear infection etc.

Surgeries with active cooling process during operation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with elective operation under general anesthesia
Sampling Method: Probability Sample
Enrollment: 2208 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-10 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
the incidence of perioperative hypothermia | from patients entered operating room to transfering to post anesthesia care units
  The core temperatures (tympanic membrane) will be measured at various time points to identify the occurence of hypothermia

SECONDARY OUTCOMES:
record the postoperative adverse events | From the day after operation to 30 days thereafter
  To identify the hypothermia related adverse events, such as cardiovascular events, wound infection, hospital stays and so on.

CONTACTS AND LOCATIONS:
Overall Officials: Yuguang Huang, doctoral, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China